CLINICAL TRIAL: NCT01559129
Title: A Phase 2, Proof-Of-Concept, Multicenter, Randomized, Double-Blind, Placebo- Controlled, Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of Pomalidomide (CC-4047) in Subjects With Systemic Sclerosis With Interstitial Lung Disease
Brief Title: Study of Pomalidomide (CC-4047) to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Effectiveness for Patients With Systemic Sclerosis With Interstitial Lung Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment was stopped early (see limitations and caveats section).
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CC-4047-SSC-001; 2010-023047-15 (EudraCT Number)
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Results first posted 2019-10-18 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Scleroderma, Systemic; Sclerosis, Systemic; Systemic Scleroderma; Systemic Sclerosis; Interstitial Lung Disease
MeSH Terms: conditions — Scleroderma, Systemic; Lung Diseases, Interstitial | interventions — pomalidomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Pomalidomide (Experimental): Participants received 1 mg pomalidomide orally once a day for 52 weeks during the treatment phase and for up to 2 years during the open-label extension phase.
  Interventions: Drug: Pomalidomide (CC-4047)

INTERVENTIONS:
Drug: Pomalidomide (CC-4047) — 1 mg orally every day for 52 weeks
  Arms: Pomalidomide
Drug: Placebo — Matching placebo capsules taken orally once a day
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety, tolerability, and efficacy of pomalidomide in the treatment of patients with systemic sclerosis with interstitial lung disease.

ELIGIBILITY:
Inclusion Criteria

* Male or females between 18 and 80 years of age (inclusive) at the time of consent.
* Diagnosis of systemic sclerosis (SSC) as defined by American College of Rheumatology (ACR) criteria.
* Onset of the first non-Raynaud's manifestation of SSC within 7 years of Screening.
* Subjects are required to meet at least one of the following 2 pulmonary-related criteria to be eligible for the study:.

  i) FVC readings ≥ 70% and ≤ 80% at Screening and Baseline (Visit 2) with a documented history of either or both of:.

A. A ≥ 5% decrease (expressed as percent predicted or in liters) in FVC in the 24-month period prior to Baseline (Visit 2) based on 3 or more assessments. Two assessments may be done during the Screening phase provided the assessments are completed at least 2 weeks apart.

B. A high resolution computed tomography (HRCT) fibrosis score > 20%.

ii) Forced vital capacity (FVC) ≥ 45% and <70% at Screening and Baseline (Visit 2) [with or without a documented pre-specified FVC decline or fibrosis score].

* FVC at Baseline (Visit 2) within 5% of the FVC measured at Screening.
* Carbon monoxide diffusing capacity (DLco) ≥ 35% and ≤ 80% of predicted value at Screening.
* Abnormalities on High-Resolution CT consistent with parenchymal changes encountered in SSc: honeycombing or reticular changes with or without ground glass.

Exclusion Criteria

* Oxygen saturation (SpO2) < 92% (room air [sea level] at rest) at Screening or Baseline.
* Known diagnosis of obstructive lung disease as defined by forced expiratory volume (FEV1)/FVC ratio < 0.7.
* Diagnosis of pulmonary arterial hypertension (PAH) requiring treatment.
* Known diagnosis of other significant respiratory disorders (e.g., asthma, tuberculosis, sarcoidosis, aspergillosis, chronic bronchitis, neoplastic disease, cystic fibrosis, etc.).
* Current clinical diagnosis of another inflammatory connective tissue disease (eg, systemic lupus erythematosus, rheumatoid arthritis, primary Sjogren's syndrome, etc.). Subjects having Sjogren's syndrome secondary to SSc are eligible.
* Pregnant or lactating females.
* History of a thromboembolic event (eg, deep vein thrombosis, thrombotic cerebrovascular or cardiovascular events).
* History or current diagnosis of peripheral neuropathy.
* Use of concomitant medication(s) which could increase the risk for developing deep vein thrombosis, including sex steroid-based contraceptives (oral, injectable or implanted) and hormone replacement therapies, if use of a low-dose aspirin regimen is contraindicated.
* Additional concomitant medications which prolong the QT/QTc interval (measure of heart's electrical cycle) during the course of the study.
* Use of any anti-coagulant or anti-thrombotic medications (other than low dose-aspirin [≤ 100 mg/day]).
* Use of any cytotoxic/immunosuppressive agent (other than prednisone ≤ 10 mg/day [mean dose] or equivalent), including but not limited to azathioprine, cyclophosphamide, methotrexate, mycophenolate and cyclosporine within 28 days (4 weeks) of Screening.
* Use of any biologic agent within 84 days (12 weeks) or 5 half-lives of Screening. In the case of rituximab, use within 168 days (24 weeks) of Screening or no recovery of CD20-positive B lymphocytes if the last dose of rituximab has been more than 24 weeks prior to Screening.
* Use of bosentan, ambrisentan, sildenafil, tadalafil and macitentan for PAH within 28 days (4 weeks) of Screening.
* Use of medications (e.g., D-penicillamine, Potaba) with putative scleroderma disease-modifying properties within 4 weeks of Screening.
* Use of melphalan within 52 weeks of Screening.
* Use of any investigational drug within 4 weeks of Screening or 5 pharmacodynamic/pharmacokinetic half-lives if known (whichever is longer).
* Smoking of cigars, pipes or cigarettes within 24 weeks of Screening.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-08-09 (Actual); Primary Completion 2016-11-03 (Actual); Study Completion 2016-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shimon Korish, MD, Study Director — Celgene Corporation
Locations (56):
- United States (20):
  - UCLA Division of Rheumatology, Los Angeles, California
  - Advances in Medicine, Rancho Mirage, California
  - Delaware Medical Care Associates, LLC, Newark, Delaware
  - Georgetown University School of Medicine, Washington D.C., District of Columbia
  - USF Health Faculty Office Building-FOB, Tampa, Florida
  - Arthritis Research and Treatment Center, Stockbridge, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - LaPorte County Institute for Clinical Research, Inc, Michigan City, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Louisiana State University, Shreveport, Louisiana
  - Boston University of Medicine BUMC, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - UMDNJ-Robert Wood Johnson Medical School Clinical Research Center, New Brunswick, New Jersey
  - North Shore-LIJ Health System-Division of Rheumatology, Great Neck, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Toledo College of Medicine, Toledo, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Monash Medical Centre, Clayton, Victoria
  - The Prince Charles Hospital, Chermside
  - The Queen Elizabeth Hospital, Woodville South
- France (3):
  - CHRU de Lille FR, Lille
  - Hopital Saint Louis, Paris
  - Groupe Hospitalier Saint Vincent de Paul, Paris
- Germany (6):
  - Kerckhoff-Klinik gGmbH, Bad Nauheim
  - Charite - Universitätsmedizin Berlin, Berlin
  - University of Erlangen-Nuremberg, Erlangen
  - Klinikum der J.W. Gothe-Universitat Frankfurt, Frankfurt
  - Rheumazentrum Ruhrgebiet, Herne
  - University Hospital of Ulm, Ulm
- Italy (7):
  - Azienda Ospedaliera Universitaria S. Martino di Genova, Genova
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale Luigi Sacco, Milan
  - IRCCS Policlinico S. Matteo di Pavia, Pavia
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Policlinico Umberto I, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
- Poland (6):
  - Centrum Miriada Prywatny Gabinet Specjalistyczny Profesora Dra Stanislawa Sierakowskiego, Bialystok
  - Szpital Uniwersytecki nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - SPSK Nr 7 Slaskiego Uniwersytetu Medycznego, Oddzial Chorob Wewnetrznych i Reumatologii, Katowice
  - Samodzielny Publiczny Szpital Kliniczny nr 1 im. prof.Tadeusza Sokolowskiego Pomorskiego UM w Szczec, Szczecin
  - Instytut Reumatologii, Klinika i Poliklinika Ukladowych Chorób Tkanki Lacznej, Warsaw
  - Akademicki Szpital Kliniczny Klinika Reumatologii i Chorob Wewnetrznych, Wroclaw
- Russia (3):
  - Institution of the Russian Academy of Medical Sciences Research Institute of Rheumatology of the Ru, Moscow
  - Penza Regional Clinical Hospital n.a. N.N. Burdenko, Penza
  - St. Petersburg State Healthcare Institution "Clinical Rheumatology Hospital # 25", Saint Petersburg
- Spain (4):
  - Hospital Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Complejo Hospitalario de Santiago, Santiago de Compostela
  - Hospital Universitario Dr. Peset, Valencia
- University Hospital Basel, Basel, Switzerland
- United Kingdom (3):
  - Chapel Allerton Hospital, Leeds
  - Royal Free Hospital, London
  - Royal Brompton Hospital - Interstitial Lung Disease Unit, London

REFERENCES:
- [Background] Hsu VM, Denton CP, Domsic RT, Furst DE, Rischmueller M, Stanislav M, Steen VD, Distler JHW, Korish S, Cooper A, Choi S, Schafer PH, Horan G, Hough DR. Pomalidomide in Patients with Interstitial Lung Disease due to Systemic Sclerosis: A Phase II, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study. J Rheumatol. 2018 Mar;45(3):405-410. doi: 10.3899/jrheum.161040. Epub 2017 Nov 1. PMID 29093152
- [Background] Hsu V, et al. A Phase 2 Study of Pomalidomide (CC-4047) to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Effectiveness in Subjects with Systemic Sclerosis with Interstitial Lung Disease. Presented at the 2016 ACR/ARHP Annual Meeting, November 11-16, 2016, Washington, DC. Abstract No. 823.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo orally once a day for 52 weeks during the treatment phase. In the open-label extension phase participants transitioned to receive 1 mg pomalidomide orally once a day for up to 2 years.
- Pomalidomide: Participants received 1 mg pomalidomide orally once a day for 52 weeks during the treatment phase and continued to receive the same treatment for up to 2 years during the open-label extension phase.
Period: Treatment Phase
Arm/Group | Placebo | Pomalidomide
Started | 12 | 11
Received Treatment | 12 | 10
Completed | 7 | 4
Not Completed | 5 | 7
Not completed — Adverse Event | 0 | 2
Not completed — Progressive Disease | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Study Terminated by Sponsor | 3 | 2
Not completed — Protocol Exclusion Criteria | 1 | 0
Not completed — Did Not Receive Study Drug | 0 | 1
Period: Open-label Extension Period
Arm/Group | Placebo | Pomalidomide
Started | 6 (One participant elected not to enter the Extension Phase.) | 2 (Two participants elected not to enter the Extension Phase.)
Completed | 0 | 0
Not Completed | 6 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Study Terminated by Sponsor | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pomalidomide | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (13.77) | 48.9 (9.84) | 46.7 (11.97)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 10 | 10 | 20
  ≥ 65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 2 | 2
  Black or African American | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islanders | 1 | 0 | 1
  White | 10 | 8 | 18
  Other | 1 | 0 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.64 (5.392) | 27.61 (9.4) | 29.19 (7.556)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen during the course of a study. A TEAE is any AE that began or worsened on or after the start of study drug through 28 days after the last dose. A treatment-related TEAE is a TEAE which was considered by the investigator to be related to study drug. The severity/intensity of AEs was assessed by the investigator as Mild (asymptomatic or mild symptoms; intervention not indicated), Moderate (symptoms cause moderate discomfort, intervention may be required), or Severe (symptoms cause severe discomfort/pain, requiring medical intervention, inability to perform daily activities). A serious AE is any AE that: - Resulted in death; - Was life-threatening; - Required inpatient hospitalization or prolongation of existing hospitalization - Resulted in persistent or significant disability/incapacity; - Was a congenital anomaly/birth defect; - Constituted an important medical event.
Time Frame: From the start of study drug to 28 days after last dose; Treatment Phase median duration of treatment was 358 and 320 days for Placebo and Pomalidomide; Extension phase median duration of treatment was 161 days and 194 days for Placebo and pomalidomide.
Population: All randomized participants who received at least one dose of the study treatment (either pomalidomide or placebo).
Measure: Number; unit: participants
Groups:
- Treatment Phase: Placebo: Participants received placebo orally once a day for 52 weeks during the treatment phase.
- Treatment Phase: Pomalidomide: Participants received 1 mg pomalidomide orally once a day for 52 weeks during the treatment phase.
- Extension Phase: Placebo/Pomalidomide: In the open-label extension phase participants received 1 mg pomalidomide orally once a day for up to 2 years.
- Extension Phase: Pomalidomide/Pomalidomide: Participants received 1 mg pomalidomide orally once a day for up to 2 years during the open-label extension phase.
Arm/Group | Treatment Phase: Placebo | Treatment Phase: Pomalidomide | Extension Phase: Placebo/Pomalidomide | Extension Phase: Pomalidomide/Pomalidomide
Number analyzed (Participants) | 12 | 10 | 6 | 2
participants
  Any TEAE | 12 | 9 | 5 | 2
  Drug-related TEAE | 8 | 6 | 3 | 1
  Severe TEAE | 1 | 4 | 0 | 0
  Serious TEAE | 1 | 4 | 0 | 1
  Serious Drug-related TEAE | 0 | 1 | 0 | 0
  TEAE Leading to Drug Interruption | 2 | 1 | 0 | 0
  TEAE Leading to Drug Withdrawal | 0 | 4 | 0 | 0
  TEAE Leading to Death | 0 | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in Percent Predicted Forced Vital Capacity (FVC) at Week 52
Description: Forced vital capacity (FVC) is a pulmonary function test and is the volume of air in the lungs that can forcibly be blown out after a full inhalation. Percent predicted values are based comparison between the participant's measured value with expected FVC for someone of the same sex, age and height (reference value). For the analysis of FVC, the baseline value was defined as the average of all values between Screening and Baseline (inclusive), and the average of Weeks 48 and 52 was treated as the Week 52 value, to reduce the total data variability at the key time points.
Time Frame: Baseline (defined as the average of all values between Screening and Baseline) and Weeks 48 and 52
Population: The Full Analysis Set (FAS) consisted of all randomized participants who received at least one dose of study drug. Participants with a Baseline value and a Week 52 were included in the analysis.
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 11 | 8
percent predicted | -2.8 (4.02) | -5.2 (5.29)

3. Primary Outcome: Change From Baseline in the Modified Rodnan Skin Score (mRSS) at Week 52/Early Termination
Description: Improvement in skin thickening is associated with improved survival and may be useful as a surrogate measurement in clinical studies. The mRSS is an assessment tool which is used to evaluate the extent and severity of the skin thickening associated with systemic sclerosis (SSc). Seventeen body areas were evaluated on a 4-point scale (0 [normal], 1 [mild], 2 [moderate]), or 3 [severe]). The total score, which is the sum of the 17 individual body assessments, can range from 0 to 51.
Time Frame: Baseline and Week 52 (or the Treatment Phase Early Termination visit)
Population: FAS participants with a Baseline value and a post-baseline value at Week 52 or Early Termination
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 11 | 10
units on a scale | -3.7 (6.99) | -2.7 (5.66)

4. Primary Outcome: Change From Baseline in University of California, Los Angeles, Scleroderma Clinical Trial Consortium Gastrointestinal Tract (UCLA SCTC GIT 2.0) Total Score at Week 52/Early Termination
Description: The UCLA SCTC GIT 2.0 is a 34-item, health-related quality of life self-administered evaluation tool, which targets gastrointestinal (GI) activity and severity in patients with SSc. Individual scales include reflux, distention/bloating, fecal soilage, diarrhea, social functioning, emotional well-being and constipation. The items are scored on a scale from 0 to 3, where 0 indicates better health and 3 indicates worse health (except for Questions 15 and 31 which are scored as 0 (better health) or 1 (worse health). The total score is calculated as the average of the first 6 scale scores (excluding constipation) which captures overall burden (severity) of SSc-associated GIT. The overall score ranges from 0 to 3, where higher scores indicate more severe symptoms.
Time Frame: Baseline and Week 52 (or Treatment Phase Early Termination visit)
Population: FAS participants with a Baseline value and a Week 52 value
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 12 | 10
units on a scale | 0.00 (0.18) | 0.1 (0.29)

5. Secondary Outcome: Change From Baseline in Percent Predicted Forced Vital Capacity Over Time
Description: Forced vital capacity (FVC) is a pulmonary function test and is the volume of air in the lungs that can forcibly be blown out after a full inhalation. Percent predicted values are based comparison between the participant's measured value with expected FVC for someone of the same sex, age and height (reference value).
Time Frame: Baseline (defined as the average of all values between Screening and Baseline) and Weeks 12, 24, 36, 64, 76, and 156
Population: FAS participants with a Baseline value and post-baseline value at the time point.
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 12 | 10
percent predicted
  Week 12: number analyzed (Participants) | 10 | 8
  Week 12 | -2.4 (3.07) | -1.8 (3.39)
  Week 24: number analyzed (Participants) | 10 | 8
  Week 24 | -1.3 (3.33) | 2.3 (12.58)
  Week 36: number analyzed (Participants) | 9 | 6
  Week 36 | -2.6 (2.48) | -4.4 (3.97)
  Week 64: number analyzed (Participants) | 6 | 2
  Week 64 | -7.0 (4.29) | -6.4 (4.49)
  Week 76: number analyzed (Participants) | 2 | 1
  Week 76 | -8.7 (10.34) | -5.2 (NA) — Could not be calculated for one participant
  Week 156: number analyzed (Participants) | 4 | 2
  Week 156 | -6.7 (6.19) | -5.9 (2.31)

6. Secondary Outcome: Change From Baseline in Modified Rodnan Skin Score Over Time
Description: Improvement in skin thickening is associated with improved survival and may be useful as a surrogate measurement in clinical studies. The mRSS is an assessment tool which is used to evaluate the extent and severity of the skin thickening associated with systemic sclerosis (SSc). Seventeen body areas were evaluated on a 4-point scale (0 [normal], 1 [mild], 2 [moderate], or 3 [severe]). The total score, which is the sum of the 17 individual body assessments, can range from 0 to 51.
Time Frame: Baseline and Weeks 12, 24, 64, 76, and 156 (or the Extension Phase Early Termination visit).
Population: FAS participants with a Baseline value and a post-baseline value at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 11 | 10
units on a scale
  Week 12: number analyzed (Participants) | 10 | 8
  Week 12 | -1.8 (3.94) | -0.3 (1.83)
  Week 24: number analyzed (Participants) | 10 | 8
  Week 24 | -3.6 (5.68) | -2.0 (3.38)
  Week 64: number analyzed (Participants) | 6 | 2
  Week 64 | -4.3 (8.36) | -4.0 (2.83)
  Week 76: number analyzed (Participants) | 2 | 1
  Week 76 | -8.5 (7.78) | -7.0 (NA) — NA = Could not be calculated for one participant
  Week 156/Early Termination: number analyzed (Participants) | 6 | 2
  Week 156/Early Termination | -3.7 (8.52) | -4.5 (3.54)

7. Secondary Outcome: Change From Baseline in UCLA SCTC GIT 2.0 Total Score Over Time
Description: The UCLA SCTC GIT 2.0 is a 34-item, health-related quality of life self-administered evaluation tool, which targets GI activity and severity in patients with SSc. Individual scales include reflux, distention/bloating, fecal soilage, diarrhea, social functioning, emotional well-being and constipation. The items are scored on a scale from 0 to 3, where 0 indicates better health and 3 indicates worse health (except for Questions 15 and 31 which are scored as 0 (better health) or 1 (worse health). The total score is calculated as the average of the first 6 scale scores (excluding constipation) which captures overall burden (severity) of SSc-associated GIT. The overall score ranges from 0 to 3, where higher scores indicate more severe symptoms.
Time Frame: Baseline and Weeks 12, 24, 64, 76, and 156 (or the Extension Phase Early Termination visit).
Population: FAS participants with a Baseline value and post-baseline value at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 12 | 10
units on a scale
  Week 12: number analyzed (Participants) | 10 | 8
  Week 12 | 0.2 (0.36) | -0.1 (0.30)
  Week 24: number analyzed (Participants) | 10 | 8
  Week 24 | 0.1 (0.23) | -0.1 (0.20)
  Week 64: number analyzed (Participants) | 6 | 2
  Week 64 | 0.0 (0.20) | 0.4 (0.01)
  Week 76: number analyzed (Participants) | 2 | 1
  Week 76 | -0.1 (0.01) | 0.5 (NA) — NA = Could not be calculated for one participant
  Week 156/Early Termination: number analyzed (Participants) | 6 | 2
  Week 156/Early Termination | 0.0 (0.14) | 0.0 (0.14)

8. Secondary Outcome: Change From Baseline in UCLA SCTC GIT 2.0 Reflux Subscale Score Over Time
Description: The UCLA SCTC GIT 2.0 is a 34-item, health-related quality of life self-administered evaluation tool, which targets GI activity and severity in patients with SSc. Individual scales include reflux, distention/bloating, fecal soilage, diarrhea, social functioning, emotional well-being and constipation. The items are scored on a scale from 0 to 3, where 0 indicates better health and 3 indicates worse health. The reflux subscale score is calculated as the average of eight reflux-related questions; the score ranges from 0 to 3, where higher scores indicate more frequent symptoms.
Time Frame: Baseline and Weeks 12, 24, 52 (or at the Treatment Phase Early Termination visit), 64, 76, and 156 (or the Extension Phase Early Termination visit).
Population: FAS participants with a Baseline value and post-baseline value at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 12 | 10
units on a scale
  Week 12: number analyzed (Participants) | 10 | 8
  Week 12 | 0.1 (0.36) | -0.1 (0.51)
  Week 24: number analyzed (Participants) | 10 | 8
  Week 24 | -0.1 (0.27) | 0.0 (0.47)
  Week 52/Early Termination | -0.1 (0.54) | 0.1 (0.38)
  Week 64: number analyzed (Participants) | 6 | 2
  Week 64 | -0.2 (0.14) | 0.2 (0.46)
  Week 76: number analyzed (Participants) | 2 | 1
  Week 76 | -0.5 (0.18) | -0.2 (NA) — NA = Could not be calculated for one participant
  Week 156/Early Termination: number analyzed (Participants) | 6 | 2
  Week 156/Early Termination | 0.0 (0.44) | 0.1 (0.28)

9. Secondary Outcome: Change From Baseline in UCLA SCTC GIT 2.0 Distension/Bloating Subscale Score Over Time
Description: The UCLA SCTC GIT 2.0 is a 34-item, health-related quality of life self-administered evaluation tool, which targets GI activity and severity in patients with SSc. Individual scales include reflux, distention/bloating, fecal soilage, diarrhea, social functioning, emotional well-being and constipation. The items are scored on a scale from 0 to 3, where 0 indicates better health and 3 indicates worse health. The distension/bloating subscale score is calculated as the average of four distension/bloating-related questions; the score ranges from 0 to 3, where higher scores indicate more frequent symptoms.
Time Frame: as for outcome 8
Population: FAS participants with a Baseline value and post-baseline value at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 12 | 10
units on a scale
  Week 12: number analyzed (Participants) | 10 | 8
  Week 12 | 0.4 (0.56) | 0.2 (1.21)
  Week 24: number analyzed (Participants) | 10 | 8
  Week 24 | 0.0 (0.53) | 0.3 (0.80)
  Week 52/Early Termination | 0.0 (0.55) | 0.2 (1.07)
  Week 64: number analyzed (Participants) | 6 | 2
  Week 64 | -0.2 (0.70) | 1.0 (1.41)
  Week 76: number analyzed (Participants) | 2 | 1
  Week 76 | 0.0 (0.00) | 3.0 (NA) — NA = Could not be calculated for one participant
  Week 156/Early Termination: number analyzed (Participants) | 6 | 2
  Week 156/Early Termination | -0.3 (0.30) | 0.9 (1.24)

10. Secondary Outcome: Change From Baseline in UCLA SCTC GIT 2.0 Fecal Soilage Subscale Score Over Time
Description: The UCLA SCTC GIT 2.0 is a 34-item, health-related quality of life self-administered evaluation tool, which targets GI activity and severity in patients with SSc. Individual scales include reflux, distention/bloating, fecal soilage, diarrhea, social functioning, emotional well-being and constipation. The items are scored on a scale from 0 to 3, where 0 indicates better health and 3 indicates worse health. The fecal soilage subscale score is calculated from one soilage question; the score ranges from 0 to 3, where higher scores indicate more frequent symptoms.
Time Frame: as for outcome 8
Population: FAS participants with a Baseline value and post-baseline value at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 12 | 10
units on a scale
  Week 12: number analyzed (Participants) | 10 | 8
  Week 12 | 0.0 (0.00) | 0.0 (0.00)
  Week 24: number analyzed (Participants) | 10 | 8
  Week 24 | 0.2 (0.42) | 0.0 (0.00)
  Week 52/Early Termination: number analyzed (Participants) | 12 | 9
  Week 52/Early Termination | 0.0 (0.00) | 0.1 (0.33)
  Week 64: number analyzed (Participants) | 6 | 2
  Week 64 | 0.2 (0.41) | 0.0 (0.00)
  Week 76: number analyzed (Participants) | 2 | 1
  Week 76 | 0.0 (0.00) | 0.0 (NA) — NA = Could not be calculated for one participant
  Week 156/Early Termination: number analyzed (Participants) | 6 | 2
  Week 156/Early Termination | 0.2 (0.41) | 0.0 (0.00)

11. Secondary Outcome: Change From Baseline in UCLA SCTC GIT 2.0 Diarrhea Subscale Score Over Time
Description: The UCLA SCTC GIT 2.0 is a 34-item, health-related quality of life self-administered evaluation tool, which targets GI activity and severity in patients with SSc. Individual scales include reflux, distention/bloating, fecal soilage, diarrhea, social functioning, emotional well-being and constipation. The diarrhea subscale score is calculated as the average of one diarrhea question about the frequency of loose stools (on a scale from 0 [none] to 3 [5-7 days/week] and one question about the presence of watery stools (scored as 0 [No] or 1 [Yes]); the score ranges from 0 to 2, where a higher score indicates more frequent symptoms.
Time Frame: as for outcome 8
Population: FAS participants with a Baseline value and post-baseline value at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 12 | 10
units on a scale
  Week 12: number analyzed (Participants) | 10 | 8
  Week 12 | 0.4 (0.57) | -0.2 (0.65)
  Week 24: number analyzed (Participants) | 10 | 8
  Week 24 | 0.1 (0.21) | -0.3 (0.46)
  Week 52/Early Termination | 0.3 (0.34) | 0.0 (0.75)
  Week 64: number analyzed (Participants) | 6 | 2
  Week 64 | 0.1 (0.38) | 0.5 (0.71)
  Week 76: number analyzed (Participants) | 2 | 1
  Week 76 | 0.0 (0.00) | -0.5 (NA) — NA = Could not be calculated for one participant
  Week 156/Early Termination: number analyzed (Participants) | 6 | 2
  Week 156/Early Termination | 0.3 (0.42) | -0.8 (0.35)

12. Secondary Outcome: Change From Baseline in UCLA SCTC GIT 2.0 Social Functioning Subscale Score Over Time
Description: The UCLA SCTC GIT 2.0 is a 34-item, health-related quality of life self-administered evaluation tool, which targets GI activity and severity in patients with SSc. Individual scales include reflux, distention/bloating, fecal soilage, diarrhea, social functioning, emotional well-being and constipation. The items are scored on a scale from 0 to 3, where 0 indicates better health and 3 indicates worse health. The social functioning subscale score is calculated as the average of six questions about how often symptoms interfered with social activities; the score ranges from 0 to 3, where higher scores indicate more frequent symptoms.
Time Frame: as for outcome 8
Population: FAS participants with a Baseline value and post-baseline value at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 11 | 10
units on a scale
  Week 12: number analyzed (Participants) | 9 | 8
  Week 12 | 0.3 (0.49) | 0.0 (0.28)
  Week 24: number analyzed (Participants) | 9 | 8
  Week 24 | 0.1 (0.30) | -0.1 (0.20)
  Week 52/Early termination | 0.0 (0.25) | 0.2 (0.45)
  Week 64: number analyzed (Participants) | 5 | 2
  Week 64 | 0.0 (0.18) | 0.3 (0.35)
  Week 76: number analyzed (Participants) | 1 | 1
  Week 76 | 0.2 (NA) — NA = Could not be calculated for one participant | 0.0 (NA) — NA = Could not be calculated for one participant
  Week 156/Early Termination: number analyzed (Participants) | 5 | 2
  Week 156/Early Termination | 0.0 (0.25) | -0.2 (0.23)

13. Secondary Outcome: Change From Baseline in UCLA SCTC GIT 2.0 Emotional Well Being Subscale Score Over Time
Description: The UCLA SCTC GIT 2.0 is a 34-item, health-related quality of life self-administered evaluation tool, which targets GI activity and severity in patients with SSc. Individual scales include reflux, distention/bloating, fecal soilage, diarrhea, social functioning, emotional well-being and constipation. The items are scored on a scale from 0 to 3, where 0 indicates better health and 3 indicates worse health. The emotional well-being subscale score is calculated as the average of nine questions regarding the impact of bowel problems on emotional status; the score ranges from 0 to 3, where higher scores indicate more frequent problems.
Time Frame: as for outcome 8
Population: FAS participants with a Baseline value and post-baseline value at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 12 | 10
units on a scale
  Week 12: number analyzed (Participants) | 10 | 8
  Week 12 | 0.2 (0.40) | -0.4 (0.80)
  Week 24: number analyzed (Participants) | 10 | 8
  Week 24 | 0.1 (0.16) | -0.3 (0.56)
  Week 52/Early Termination | 0.1 (0.25) | -0.1 (0.42)
  Week 64: number analyzed (Participants) | 6 | 2
  Week 64 | 0.0 (0.36) | 0.2 (0.00)
  Week 76: number analyzed (Participants) | 2 | 1
  Week 76 | 0.0 (0.00) | 0.3 (NA) — NA = Could not be calculated for one participant
  Week 156/Early Termination: number analyzed (Participants) | 6 | 2
  Week 156/Early Termination | -0.1 (0.15) | 0.0 (0.00)

14. Secondary Outcome: Change From Baseline in UCLA SCTC GIT 2.0 Constipation Subscale Score Over Time
Description: The UCLA SCTC GIT 2.0 is a 34-item, health-related quality of life self-administered evaluation tool, which targets GI activity and severity in patients with SSc. Individual scales include reflux, distention/bloating, fecal soilage, diarrhea, social functioning, emotional well-being and constipation. The items are scored on a scale from 0 to 3, where 0 indicates better health and 3 indicates worse health. The constipation subscale score is calculated as the average of three questions regarding the frequency of constipation (scored from 0 [no days] to 3 [5-7 days/week] and one question about the presence of stools becoming harder (scored as 0 [No] or 1 [Yes]); the score ranges from 0 to 2.5, where higher scores indicate more frequent symptoms.
Time Frame: as for outcome 8
Population: FAS participants with a Baseline value and post-baseline value at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 12 | 10
units on a scale
  Week 12: number analyzed (Participants) | 10 | 8
  Week 12 | -0.1 (0.36) | 0.2 (0.98)
  Week 24: number analyzed (Participants) | 10 | 8
  Week 24 | -0.2 (0.31) | 0.3 (0.81)
  Week 52/Early Termination | 0.0 (0.25) | 0.3 (0.51)
  Week 64: number analyzed (Participants) | 6 | 2
  Week 64 | 0.0 (0.60) | 0.1 (0.18)
  Week 76: number analyzed (Participants) | 2 | 1
  Week 76 | 0.0 (0.00) | 0.0 (NA) — NA = Could not be calculated for one participant
  Week 156/Early Termination: number analyzed (Participants) | 6 | 2
  Week 156/Early Termination | -0.2 (0.20) | 0.1 (0.18)

15. Secondary Outcome: Change From Baseline in Dyspnea Functional Impairment at Week 12
Description: The Transition Dyspnea Index (TDI) provides interview-based measurements of breathlessness related to activities of daily living. The TDI is an evaluative instrument that includes specific criteria for each of three components (functional impairment, magnitude of task and magnitude of effort) to measure changes from a baseline state. Changes in dyspnea functional impairment were assessed on a scale from Major Deterioration (formerly working but had to stop working and abandoned usual activities due to shortness of breath) to Major Improvement (able to return to work at former pace and return to full activities with only mild restriction due to improvement of shortness of breath). Further impairment for other reasons includes participants who gave up or reduced work or other activities for reasons other than shortness of breath.
Time Frame: Week 12
Population: FAS participants with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 10 | 7
Participants
  Major deterioration | 0 | 0
  Moderate deterioration | 1 | 1
  Minor deterioration | 0 | 1
  No change | 7 | 3
  Minor improvement | 2 | 1
  Moderate improvement | 0 | 0
  Major improvement | 0 | 0
  Further impairment for other reasons | 0 | 1

16. Secondary Outcome: Change From Baseline in Dyspnea Functional Impairment at Week 24
Description: as for outcome 15
Time Frame: Week 24
Population: FAS participants with available data
Measure: Number; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 10 | 7
Participants
  Major deterioration | 1 | 0
  Moderate deterioration | 0 | 2
  Minor deterioration | 1 | 1
  No change | 4 | 2
  Minor improvement | 3 | 1
  Moderate improvement | 1 | 0
  Major improvement | 0 | 0
  Further impairment for other reasons | 0 | 1

17. Secondary Outcome: Change From Baseline in Dyspnea Functional Impairment at Week 52/Early Termination
Description: as for outcome 15
Time Frame: Week 52 or at the Treatment Phase Early Termination visit
Population: FAS participants with available data
Measure: Number; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 12 | 10
Participants
  Major deterioration | 0 | 0
  Moderate deterioration | 0 | 4
  Minor deterioration | 1 | 1
  No change | 8 | 4
  Minor improvement | 3 | 1
  Moderate improvement | 0 | 0
  Major improvement | 0 | 0
  Further impairment for other reasons | 0 | 0

18. Secondary Outcome: Change From Baseline in Dyspnea Functional Impairment at Week 64
Description: as for outcome 15
Time Frame: Week 64
Population: FAS participants with available data
Measure: Number; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 6 | 2
Participants
  Major deterioration | 0 | 1
  Moderate deterioration | 0 | 1
  Minor deterioration | 1 | 0
  No change | 4 | 0
  Minor improvement | 1 | 0
  Moderate improvement | 0 | 0
  Major improvement | 0 | 0
  Further impairment for other reasons | 0 | 0

19. Secondary Outcome: Change From Baseline in Dyspnea Functional Impairment at Week 76
Description: as for outcome 15
Time Frame: Week 76
Population: FAS participants with available data
Measure: Number; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 2 | 1
Participants
  Major deterioration | 0 | 0
  Moderate deterioration | 0 | 1
  Minor deterioration | 1 | 0
  No change | 0 | 0
  Minor improvement | 1 | 0
  Moderate improvement | 0 | 0
  Major improvement | 0 | 0
  Further impairment for other reasons | 0 | 0

20. Secondary Outcome: Change From Baseline in Dyspnea Functional Impairment at Week 156/Early Termination
Description: as for outcome 15
Time Frame: Week 156 or the Extension Phase Early Termination visit
Population: FAS participants with available data
Measure: Number; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 6 | 2
Participants
  Major deterioration | 0 | 0
  Moderate deterioration | 0 | 1
  Minor deterioration | 2 | 1
  No change | 2 | 0
  Minor improvement | 1 | 0
  Moderate improvement | 1 | 0
  Major improvement | 0 | 0
  Further impairment for other reasons | 0 | 0

21. Secondary Outcome: Change From Baseline in Dyspnea Magnitude of Task at Week 12
Description: The Transition Dyspnea Index (TDI) provides interview-based measurements of breathlessness related to activities of daily living. The TDI is an evaluative instrument that includes specific criteria for each of three components (functional impairment, magnitude of task and magnitude of effort) to measure changes from a baseline state. At Baseline magnitude of task was assessed on a scale from Grade 0 (becomes short of breath at rest, while sitting or lying) to Grade 4 (becomes short of breath only with extraordinary activity such as running or carrying very heavy loads). Changes in dyspnea magnitude of task were assessed on a scale from Major Deterioration (deteriorated ≥ 2 grades from Baseline) to Major Improvement (Improved ≥ 2 grades from Baseline). Further impairment for other reasons includes participants with reduced exertion capacity for reasons other than shortness of breath, for example musculoskeletal problems or chest pain.
Time Frame: Week 12
Population: FAS participants with available data
Measure: Number; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 10 | 7
Participants
  Major deterioration | 0 | 0
  Moderate deterioration | 0 | 0
  Minor deterioration | 2 | 1
  No change | 5 | 5
  Minor improvement | 3 | 1
  Moderate improvement | 0 | 0
  Major improvement | 0 | 0
  Further impairment for other reasons | 0 | 0

22. Secondary Outcome: Change From Baseline in Dyspnea Magnitude of Task at Week 24
Description: as for outcome 21
Time Frame: Week 24
Population: FAS participants with available data
Measure: Number; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 10 | 7
Participants
  Major deterioration | 0 | 0
  Moderate deterioration | 1 | 1
  Minor deterioration | 2 | 1
  No change | 5 | 2
  Minor improvement | 2 | 3
  Moderate improvement | 0 | 0
  Major improvement | 0 | 0
  Further impairment for other reasons | 0 | 0

23. Secondary Outcome: Change From Baseline in Dyspnea Magnitude of Task at Week 52/Early Termination
Description: as for outcome 21
Time Frame: Week 52 or at the Treatment Phase Early Termination visit
Population: FAS participants with available data
Measure: Number; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 12 | 10
Participants
  Major deterioration | 0 | 0
  Moderate deterioration | 0 | 3
  Minor deterioration | 1 | 1
  No change | 8 | 6
  Minor improvement | 2 | 0
  Moderate improvement | 0 | 0
  Major improvement | 1 | 0
  Further impairment for other reasons | 0 | 0

24. Secondary Outcome: Change From Baseline in Dyspnea Magnitude of Task at Week 64
Description: as for outcome 21
Time Frame: Week 64
Population: FAS participants with available data
Measure: Number; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 6 | 2
Participants
  Major deterioration | 0 | 1
  Moderate deterioration | 0 | 0
  Minor deterioration | 2 | 0
  No change | 3 | 0
  Minor improvement | 1 | 1
  Moderate improvement | 0 | 0
  Major improvement | 0 | 0
  Further impairment for other reasons | 0 | 0

25. Secondary Outcome: Change From Baseline in Dyspnea Magnitude of Task at Week 76
Description: as for outcome 21
Time Frame: Week 76
Population: FAS participants with available data
Measure: Number; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 2 | 1
Participants
  Major deterioration | 0 | 0
  Moderate deterioration | 0 | 0
  Minor deterioration | 1 | 0
  No change | 1 | 0
  Minor improvement | 0 | 1
  Moderate improvement | 0 | 0
  Major improvement | 0 | 0
  Further impairment for other reasons | 0 | 0

26. Secondary Outcome: Change From Baseline in Dyspnea Magnitude of Task at Week 156/Early Termination
Description: The Transition Dyspnea Index (TDI) provides interview-based measurements of breathlessness related to activities of daily living. The TDI is an evaluative instrument that includes specific criteria for each of three components (functional impairment, magnitude of task and magnitude of effort) to measure changes from a baseline state. At Baseline magnitude of task was assessed on a scale from Grade 0 (becomes short of breath at rest, while sitting or lying) to Grade 4 (becomes short of breath only with extraordinary activity such as running or carry very heavy loads). Changes in dyspnea magnitude of task were assessed on a scale from Major Deterioration (deteriorated ≥ 2 grades from Baseline) to Major Improvement (Improved ≥ 2 grades from Baseline). Further impairment for other reasons includes participants with reduced exertion capacity for reasons other than shortness of breath, for example musculoskeletal problems or chest pain.
Time Frame: Week 156 or the Extension Phase Early Termination visit
Population: FAS participants with available data
Measure: Number; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 6 | 2
Participants
  Major deterioration | 0 | 0
  Moderate deterioration | 1 | 0
  Minor deterioration | 1 | 1
  No change | 2 | 0
  Minor improvement | 2 | 1
  Moderate improvement | 0 | 0
  Major improvement | 0 | 0
  Further impairment for other reasons | 0 | 0

27. Secondary Outcome: Change From Baseline in Dyspnea Magnitude of Effort at Week 12
Description: The Transition Dyspnea Index (TDI) provides interview-based measurements of breathlessness related to activities of daily living. The TDI is an evaluative instrument that includes specific criteria for each of three components (functional impairment, magnitude of task and magnitude of effort) to measure changes from a baseline state. At Baseline magnitude of task was assessed on a scale from Grade 0 (becomes short of breath at rest, while sitting or lying) to Grade 4 (becomes short of breath only with greatest imaginable effort). Changes in dyspnea magnitude of task were assessed on a scale from Major Deterioration (severe decrease in effort from Baseline to avoid shortness of breath, activities take 50-100% longer to complete) to Major Improvement (able to do things with much greater effort than previously with few, if any, pauses). Further impairment for other reasons includes participants with reduced exertion capacity for reasons other than shortness of breath.
Time Frame: Week 12
Population: FAS participants with available data
Measure: Number; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 10 | 7
Participants
  Major deterioration | 0 | 0
  Moderate deterioration | 1 | 0
  Minor deterioration | 2 | 2
  No change | 4 | 4
  Minor improvement | 2 | 1
  Moderate improvement | 1 | 0
  Major improvement | 0 | 0
  Further impairment for other reasons | 0 | 0

28. Secondary Outcome: Change From Baseline in Dyspnea Magnitude of Effort at Week 24
Description: as for outcome 27
Time Frame: Week 24
Population: FAS participants with available data
Measure: Number; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 10 | 7
Participants
  Major deterioration | 1 | 1
  Moderate deterioration | 0 | 1
  Minor deterioration | 1 | 0
  No change | 4 | 3
  Minor improvement | 3 | 2
  Moderate improvement | 1 | 0
  Major improvement | 0 | 0
  Further impairment for other reasons | 0 | 0

29. Secondary Outcome: Change From Baseline in Dyspnea Magnitude of Effort at Week 52/Early Termination
Description: as for outcome 27
Time Frame: Week 52 or at the Treatment Phase Early Termination visit
Population: FAS participants with available data
Measure: Number; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 12 | 10
Participants
  Major deterioration | 0 | 0
  Moderate deterioration | 0 | 3
  Minor deterioration | 1 | 1
  No change | 7 | 6
  Minor improvement | 3 | 0
  Moderate improvement | 1 | 0
  Major improvement | 0 | 0
  Further impairment for other reasons | 0 | 0

30. Secondary Outcome: Change From Baseline in Dyspnea Magnitude of Effort at Week 64
Description: as for outcome 27
Time Frame: Week 64
Population: FAS participants with available data
Measure: Number; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 6 | 2
Participants
  Major deterioration | 0 | 1
  Moderate deterioration | 0 | 0
  Minor deterioration | 3 | 0
  No change | 2 | 1
  Minor improvement | 1 | 0
  Moderate improvement | 0 | 0
  Major improvement | 0 | 0
  Further impairment for other reasons | 0 | 0

31. Secondary Outcome: Change From Baseline in Dyspnea Magnitude of Effort at Week 76
Description: as for outcome 27
Time Frame: Week 76
Population: FAS participants with available data
Measure: Number; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 2 | 1
Participants
  Major deterioration | 0 | 0
  Moderate deterioration | 0 | 0
  Minor deterioration | 1 | 0
  No change | 0 | 1
  Minor improvement | 1 | 0
  Moderate improvement | 0 | 0
  Major improvement | 0 | 0
  Further impairment for other reasons | 0 | 0

32. Secondary Outcome: Change From Baseline in Dyspnea Magnitude of Effort at Week 156/Early Termination
Description: as for outcome 27
Time Frame: Week 156 or at the Extension Phase Early Termination visit
Population: FAS participants with available data
Measure: Number; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 6 | 2
Participants
  Major deterioration | 0 | 0
  Moderate deterioration | 1 | 0
  Minor deterioration | 2 | 1
  No change | 2 | 1
  Minor improvement | 1 | 0
  Moderate improvement | 0 | 0
  Major improvement | 0 | 0
  Further impairment for other reasons | 0 | 0

33. Secondary Outcome: Oxygen Saturation Over Time
Description: Oxygen saturation was measured by pulse oximetry.
Time Frame: as for outcome 8
Population: FAS participants with a value at each time point.
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 12 | 9
percent saturation
  Baseline | 97.5 (2.07) | 96.8 (1.92)
  Week 12: number analyzed (Participants) | 10 | 8
  Week 12 | 97.1 (2.18) | 97.4 (1.51)
  Week 24: number analyzed (Participants) | 10 | 8
  Week 24 | 97.6 (1.65) | 96.5 (4.31)
  Week 52/Early Termination | 96.8 (2.18) | 96.8 (1.86)
  Week 64: number analyzed (Participants) | 6 | 2
  Week 64 | 96.3 (2.94) | 94.0 (2.83)
  Week 76: number analyzed (Participants) | 2 | 1
  Week 76 | 98.5 (0.71) | 97.0 (NA) — NA = Could not be calculated for one participant
  Week 156/Early Termination: number analyzed (Participants) | 6 | 2
  Week 156/Early Termination | 95.8 (5.12) | 97.5 (0.71)

34. Secondary Outcome: Pharmacokinetic Parameters of Pomalidomide in Plasma
Description: Pharmacokinetic (PK) analyses were not conducted as there were too few participants with available data.
Time Frame: Day 1 and week 4 pre-dose and up to 24 hours post-dose.
Population: PK analyses were not conducted as there were too few participants with available data. No data was analyzed.
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the start of study drug to 28 days after last dose; Treatment Phase median duration of treatment was 358 and 320 days for Placebo and Pomalidomide; Extension phase median duration of treatment was 161 days and 194 days for Placebo and Pomalidomide.
Arm/Group | Treatment Phase: Placebo | Treatment Phase: Pomalidomide | Extension Phase: Placebo/Pomalidomide | Extension Phase: Pomalidomide/Pomalidomide
Serious Adverse Events (participants affected / at risk) | 1/12 | 4/10 | 0/6 | 1/2
Other Adverse Events (participants affected / at risk) | 12/12 | 9/10 | 5/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Phase: Placebo (N=12) | Treatment Phase: Pomalidomide (N=10) | Extension Phase: Placebo/Pomalidomide (N=6) | Extension Phase: Pomalidomide/Pomalidomide (N=2)
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Phase: Placebo (N=12) | Treatment Phase: Pomalidomide (N=10) | Extension Phase: Placebo/Pomalidomide (N=6) | Extension Phase: Pomalidomide/Pomalidomide (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mucous stools (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Device breakage (General disorders) | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 0 | 0
Pain (General disorders) | 1 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 2 | 0
Laryngitis viral (Infections and infestations) | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Blood iron decreased (Investigations) | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 1 | 1 | 0 | 0
Heart rate increased (Investigations) | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Digital ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Menopause (Social circumstances) | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Based upon interim analysis data, the study did not meet its primary endpoints for subjects who had completed blinded treatment. The IDMC recommended the study be stopped due to lack of efficacy and the sponsor agreed with this recommendation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.